CLINICAL TRIAL: NCT01800669
Title: Computer-Supported Management of Medical-Legal Issues Impacting Child Health
Acronym: CHICA-MLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1R01HS020640-01A1 (AHRQ)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Legal Rights; Medicolegal Aspects
Keywords: Computer based clinical decision support; medical legal partnership; child; pediatrics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Use of the complete CHICA MLP module in routine clinical care. The MLP module screens families for medical-legal issues, alerts the physician to there presences and provides guidance and referral materials to help the physician resolve the issues.
  Interventions: Other: CHICA MLP Module
- Control (Active Comparator): CHICA without the MLP module. This version includes a module that screens families for medical-legal issue but does not provide additional guidance or referrals to resolve them.
  Interventions: Other: CHICA without the MLP module

INTERVENTIONS:
Other: CHICA MLP Module — The MLP module screens families for medical-legal issues, alerts the physician to there presences and provides guidance and referral materials to help the physician resolve the issues.
  Arms: Intervention
Other: CHICA without the MLP module — Clinics in the control group will have the CHICA system, but without the MLP module. It will screen for medical-legal issues but will not provide additional guidance and referrals to help resolve them.
  Arms: Control

SUMMARY:
The investigators hypothesize that by adding a patient screening and physician alerting module to a computer-based decision support system, the investigators can improve the detection and management of legal issues that may affect children's health. this randomized controlled trial will place the module in two clinics using the CHICA decision support system and compare the rate of detection and resolution of medical-legal issues in those clinics compared to two clinics using the CHICA system without the medical-legal module.

DETAILED DESCRIPTION:
Social determinants of health are the circumstances in which people are born, live, work and age; as well as the systems that are put in place to deal with illness and disability. Dramatic differences in health are closely related to degrees of social and economic disadvantage. For example, poverty-induced hardships such as food insecurity, utility shut-offs and substandard housing all have the potential to negatively impact health. In the United States, there exist many laws and policies designed to address such issues. For example, the Supplemental Nutrition Assistance Program (SNAP) seeks to address food insecurity by providing a means for financially eligible recipients to access nutritious food. When an individual is wrongly denied SNAP benefits, legal remedies are available. Access to legal aid, much like access to nutritious food, is often limited by social and economic disadvantage. It has been demonstrated that most legal problems experienced by low-income individuals remain unresolved, with fewer than one in five being addressed with the help of a lawyer.

A child's health status may be negatively affected when he or she does not receive the benefit of laws designed to address such social determinates of health. Unhealthy housing may lead to an increased risk of preventable injury or, in the case of dangerous molds, asthma. An excessively cold environment brought on by a utility shut-off may also trigger childhood asthma, or result in a family's decision to trade-off food for heat. Poor nutrition may contribute to any number of deficiencies impacting a child's health. Laws addressing such issues include those that require landlords to mitigate dangerous rental housing conditions, those that protect access to utilities in certain circumstances, and those that protect against unlawful denials of food-benefit programs.

Medical-legal Partnerships bring health care providers together with lawyers to address social and legal needs, such as those described above, which may result in poor health outcomes. Such partnerships across the nation provide direct legal advice and assistance to patients, create internal systems that improve health care delivery, and promote change at a policy level beyond discrete systems. This study has been designed to expand upon the current medical-legal partnership concept and mitigate health disparities by creating an innovative system that dramatically increases the identification of medical-legal issues in pediatric clinics, improves the delivery of appropriate physician counseling and streamlines access to legal resources when legal remedies are needed.

The investigators propose to intelligently insert a medical-legal issue screening tool and tailored decision support protocol into the regular health care delivery process of our existing computerized clinical decision support system (CDSS), the Child Health Improvement through Computer Automation (CHICA) system. In short, a series of screening questions regarding common legal issues that have the potential to negatively impact child health will be included on a pre-screener form for all patients ≤36 months of age. This form will be printed on paper and completed by the presenting caregiver in the waiting room. Answers to the questions will then be scanned into the CHICA system prior to the physician encounter and analyzed along with previously existing medical record information to generate the content for a tailored physician worksheet and handouts. Together, these documents will help guide physicians through the process of confirming identified medical-legal issues and providing the most appropriate interventions in terms of education and/or referrals to a medical-legal expert. This process as a whole will help physicians to accurately identify such issues and immediately address them in an appropriate and sensitive way.

The investigators hypothesize that our innovative use of the CHICA computerized decision support system to identify and address medical-legal issues in a consistent, appropriate and effective way will help diminish the barriers that physicians often cite when questioned about identifying medical-legal issues and taking steps to help address them. For example, the investigators anticipate that our utilization of waiting room time to administer the initial pre-screener questions will help minimize concerns about time constraints, and CHICA's generation of highly-tailored worksheets that direct physicians through the process of dealing with positive screens will help address physician concerns about lack of education or experience with medical-legal issues.

To summarize, the investigators intend first to expand and modify the CHICA system to assist pediatricians with the identification and management of four common medical-legal problems (homelessness, unsafe rental home conditions, inadequate access to necessary utilities and food insecurity) that have the potential to adversely impact child health (AIM 1). The investigators will then evaluate the effect of the CHICA medical-legal module on the identification and mitigation of medical-legal problems in four pediatric practices by evaluating rates of medical-legal issue identification via pre/post chart abstraction, and evaluating actions taken by physicians and patient caregivers (as reported in caregiver interviews) to mitigate identified medical-legal issues (AIM 2). Next, the investigators will evaluate physician and patient caregiver satisfaction with the CHICA medical-legal module by evaluating physician comfort with medical-legal issue identification and acceptance of the CHICA medical-legal module via physician survey, and evaluating patient caregiver perceptions (as reported in caregiver interviews) about physicians' handling of medical-legal issues and the CHICA medical-legal module process (AIM 3). Lastly, the investigators will evaluate the impact of the CHICA medical-legal module on healthcare utilization by comparing the overall utilization of Medicaid patients in our intervention population to Medicaid patients in our control population over the course of 18 months (AIM 4).

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 2 years
* Attending one of the intervention or control clinics in Indianapolis

Exclusion Criteria:

* Inability to complete study materials (provided in English and Spanish)

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 582 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rates of detection of medical-legal issues | 1 year
  Rates of detection of medical-legal issues among families of children attending intervention or control clinics. Outcome will be assessed by chart abstraction before and one year after onset of the intervention.

SECONDARY OUTCOMES:
Rates of resolution of medical-legal issues. | 1 year
  Rates of resolution of medical-legal issues among families with medical-legal issues will be assessed by face-to-face interviews of care givers seeking healthcare for their children in one of the study clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Gilbert, JD, MPH, Principal Investigator — Indiana University
Locations (1):
- Wishard/Eskenazi Hospital Clinics, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Gilbert AL, Downs SM. Medical legal partnership and health informatics impacting child health: Interprofessional innovations. J Interprof Care. 2015;29(6):564-9. doi: 10.3109/13561820.2015.1029066. Epub 2015 Jun 29. PMID 26120893
- See also: Research Group Carrying out the Study — http://www.ichsr.org/